CLINICAL TRIAL: NCT03003104
Title: A Randomized, Double-Blind, Vehicle Controlled Study To Evaluate The Safety, Tolerability, And Efficacy Of DMT210 Gel In Adult Patients With Moderate To Severe Acne Rosacea
Brief Title: DMT210 Topical Gel in the Treatment of Acne Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermata Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMT210-003
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Acne Rosacea
Keywords: Skin diseases; rosacea
MeSH Terms: conditions — Rosacea; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMT210 Topical Gel (Experimental): DMT210 Topical Gel 5% applied to the face twice daily for 12 weeks
  Interventions: Drug: DMT210 Topical Gel 5%
- Vehicle Control (Placebo Comparator): Topical Gel vehicle applied to the face twice daily for 12 weeks
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Drug: DMT210 Topical Gel 5%
  Arms: DMT210 Topical Gel
Other: Vehicle Control
  Arms: Vehicle Control

SUMMARY:
The study evaluates the safety, tolerability, and efficacy of DMT210 Gel, 5% when applied twice daily for 12 weeks in adult patients with moderate to severe acne rosacea. Half of participants will receive DMT210 Gel while the other half will receive vehicle control.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or non-pregnant female at least 18 years of age.
* Clinical diagnosis of moderate to severe facial rosacea as determined by Investigator's Global Assessment (IGA) at Randomization
* Patient has at least ten inflammatory lesions of rosacea on the face at Randomization
* Patient is willing to apply the Investigational Product as directed
* Patient is willing and able to comply with the protocol

Exclusion Criteria:

* Patient is pregnant or planning to become pregnant
* Patient is taking a topical therapy which may affect the patient's rosacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by Inflammatory lesion counts | 12 weeks
  Inflammatory lesion counts
Efficacy as measured by Investigator Global Assessment (IGA) | 12 weeks
  Investigator Global Assessment (IGA)
Efficacy as measured by 5-point Clinical Erythema Assessment (CEA) | 12 weeks
  5-point Clinical Erythema Assessment (CEA)
Efficacy as measured by 5-point Patient Severity Assessment of Erythema (PSA) | 12 weeks
  5-point Patient Severity Assessment of Erythema (PSA)

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 12 weeks
  Incidence of adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Dermata Investigational Site, San Diego, California
  - Dermata Investigational Site, Miami, Florida
  - Dermata Investigational Site, Fridley, Minnesota
  - Dermata Investigational Site, Omaha, Nebraska
  - Dermata Investigational Site, High Point, North Carolina
  - Dermata Investigational Site, Broomall, Pennsylvania
  - Dermata Investigational Site, Nashville, Tennessee
  - Dermata Investigational Site, Austin, Texas
  - Dermata Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No